CLINICAL TRIAL: NCT07395011
Title: The Effectiveness of Dynamic Neuromuscular Stabilization (DNS) Exercises Compared to Localized Exercises and Standard Care on Pain Intensity, Neck Dysfunction, and Upper Cervical Range of Motion in Patients With Chronic Neck Pain: A Pilot Randomized Controlled Trial (RCT)
Acronym: DYNEX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hochschule Osnabruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WiSo_BA_PTB_WiSe25-26_1_1
Record Dates: First submitted 2026-01-31; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Neck Pain; Neck Pain Musculoskeletal; Chronic Neck Pain; Neck Disease; Neck Disability
MeSH Terms: conditions — Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DNS_Group (Experimental)
  Interventions: Other: Dynamic Neuromuscular Stabilization (DNS) Exercises
- Local_Exercise (Experimental)
  Interventions: Other: Local Exercises
- Usual_Care (Experimental)
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Dynamic Neuromuscular Stabilization (DNS) Exercises — Dynamic Neuromuscular Stabilization (DNS) is a physiotherapy approach based on developmental kinesiology. It uses specific postural and breathing exercises to restore spinal stability, improve motor control, and enhance cervical function under physiotherapist supervision.
  Arms: DNS_Group
Other: Local Exercises — Localized neck exercises target deep and superficial cervical muscles through specific strengthening, motor control, and stabilization drills. The program includes chin tucks, resisted movements, and scapular stabilization, supervised by a physiotherapist to improve pain, function, and coordination.
  Arms: Local_Exercise
Other: Usual Care — Usual care includes standard physiotherapy for chronic neck pain: patient education, manual therapy, heat application, and general stretching or mobility exercises. Treatment follows typical clinical practice and is adjusted to individual needs.
  Arms: Usual_Care

SUMMARY:
Many people experience long-lasting neck pain, which can affect daily life, work, and overall well-being. This study aims to find out which type of exercise program is most effective in reducing neck pain, improving neck movement, and making daily activities easier.

What Is Being Studied?:

The study compares three different types of treatment:

DNS Exercises (Dynamic Neuromuscular Stabilization):

Whole-body exercises focusing on posture, breathing, and core stability.

Localized Neck Exercises:

Targeted exercises for the neck and shoulder muscles.

Standard Care:

Usual physiotherapy treatment commonly provided in clinical practice.

Study Procedures:

Participants are randomly assigned to one of the three groups. Each participant receives individual exercise instruction from a physiotherapist.

Participants are also given simple home exercises to perform on their own. The study lasts for about 12 weeks.

What Will Be Measured?:

At the beginning, during, and at the end of the study, the following will be assessed:

Neck pain intensity (pain scale) Neck range of motion How much the pain affects daily life and activities

Possible Benefits:

Participants may experience:

Less neck pain Improved neck mobility Better overall body awareness Even if not every participant notices improvement, taking part will help researchers improve future treatment options for chronic neck pain.

Risks:

No major risks are expected. All exercises are supervised by qualified physiotherapists and adjusted to each participant's abilities.

Participation can be stopped at any time if discomfort or pain occurs.

Voluntary Participation and Data Privacy:

Participation is completely voluntary. All personal data will be kept confidential and analyzed anonymously for research purposes only.

Participants may withdraw from the study at any time without any disadvantages.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 50 years of age. This ensures a homogeneous population that in-cludes both young adults and middle-aged individuals.
* have suffered from neck pain continuously for at least 12 weeks, as described by the International Association for the Study of Pain (IASP)
* have current neck pain greater than 40 on the Numeric Rating Scale (NRS) (on a scale of 0 to 100).
* have an NDI score of over 10 points.

Exclusion Criteria: -

* Cancer
* Patients with existing or previous fractures in the cervical spine
* Patients who have undergone surgery on the cervical spine
* Patients who, in addition to neck pain, also have or have had dizziness or balance disorders
* People with osteoporosis
* Fibromyalgia
* People with diagnosed rheumatoid arthritis
* People with red flags identified during a thorough physical examination
* Patients with neurological deficits identified during a thorough physical examination
* Participants who have undergone physiotherapy within the last 3 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Ratic Scale | From enrollment to the end of treatment at 12 weeks

SECONDARY OUTCOMES:
Neck Disability Index | From enrollment to the end of treatment at 12 weeks
Flexio Rotation Test | From enrollment to the end of treatment at 12 weeks
Fear-Avoidance Beliefs Questionnaire | From enrollment to the end of treatment at 12 weeks